CLINICAL TRIAL: NCT06396546
Title: 'Glycogen Storage Diseases (GSDs) in Indian Children- Establishing an Indian GSD (I-GSD) Registry'.
Acronym: I-GSD
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-GSD-01
Record Dates: First submitted 2024-04-13; First posted 2024-05-02 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-04

CONDITIONS: Glycogen Storage Diseases
MeSH Terms: conditions — Glycogen Storage Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glycogen storage disorders (GSD) are a class of inborn metabolic abnormalities characterized by enzymatic defects in glycogen production or breakdown and are one of commonest metabolic disorders of the childhood. Their pathogenesis mostly involves the liver and muscles and can range in severity from minor disorders with a typical lifespan to those that are fatal in infancy. Different GSDs, such as type 0a, I, III (most common type), IV, VI, IX, and XI (based on specific gene variants) are now referred to as hepatic GSDs involving liver (+ muscle). GSDs show clinically in a wide range of ways, and they have typically been identified by combining clinical symptoms, biochemical data, and pathological findings. But due to lack of multicentre evaluation, there is persistent scarcity of data with regard to the overall spectrum of genetic defects in Indian children presenting with GSD, their natural course and genotype-phenotype correlation. Also, there is limited data on common genetic variations in Indian population causing hepatic glycogen storage diseases.

An Indian GSD registry is needed to describe the spectrum, natural course, genotype-phenotype correlation, outcome and response to medical therapy in Indian children with GSDs. The study would be the first to extensively describe the genotype of Indian children with GSD and their natural course. Being a multicentric study, the results generated would therefore be applicable to the whole of the country. Understanding the prevalent genotypes in Indian population and their related phenotype would help both the individual management decisions of these patients and further policy making for their diagnosis and treatment. Results from this study could thus guide appropriate decision making based on outcome and help choose the modality of treatment for the individual patient - medical, or liver transplantation.

DETAILED DESCRIPTION:
* Primary objective:
* To describe the clinical presentation and outcome of genetically defined cases of pediatric hepatic glycogen storage diseases (GSD) patients.
* Study population: Genetically confirmed cases of hepatic GSDs will be enrolled from all the participating centres.
* Study design: Multicentric retrospective study (with concomitant long term prospective data collection)
* Study period: The study will be an ongoing effort with aim to continuosly expand the participation. Retrospective data collection (of previous data), analysis and drafting of manuscript would be completed between May 2024 to April 2025. New centers willing to join the consortium will be asked to submit their data as on the date of joining. Retrospective follow up data may be asked from the participating centres every every 6 months-1 year. Also, we would continue prospective data collection of newer GSD patients at the collaborating centres.

ELIGIBILITY:
Inclusion Criteria:

* Children <18 years of age (at presentation) with genetically proven (homozygous or compound heterozygous mutations) hepatic glycogen storage diseases

  1. types 0a/GYS2 gene, I/G6PC or SLC37A4 gene variants, III/ AGL gene variants, IV/ GBE1 gene variants, VI/ PYGL gene variants, IX/ PHKA2, PHKB or PHKG2 gene variants and XI/ GLUT2/SLC2A2 gene variants.

     Exclusion Criteria:

     -
* Clinical, biochemical and histological evidence of GSDs without a confirmatory genetic sequencing report.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Genetically confirmed cases of hepatic GSDs will be enrolled from all the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate clinical presentation and outcome (long term native liver or post liver transplant survival etc) of genetically defined cases of Indian pediatric hepatic glycogen storage diseases (GSD) patients. | 5 years
  Clinical presentation defined as symptomatology, biochemical and genetic features etc.

SECONDARY OUTCOMES:
Various types of genetic variations (missense, nonsense, frameshift etc) in Indian children with GSD. | Day 0
Association between specific genetic variations (genotype) and the resulting clinical disease expression (phenotype) in Indian children with various types of hepatic GSDs. | 5 years
To evaluate the complications and outcome after liver transplantation in Indian children with various types of hepatic GSDs. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Vikrant Sood, DM, Study Director — Institute of Liver & Biliary Sciences
Locations (3):
- India (3):
  - Government Medical College, Thiruvananthapuram, Kerala
  - KEM Hospital, Pune, Maharashtra
  - Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Undecided